CLINICAL TRIAL: NCT01942304
Title: Prospective Evaluation of Anorganic Bovine Bone Mineral Versus Calcium Phosphosilicate Alloplastic Bone Putty in Direct Sinus Augmentation: a Spilt-mouth Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: NovaBone Products, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1308M40681
Record Dates: First submitted 2013-09-10; First posted 2013-09-13 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Sinus Floor Augmentation; Maxillary Sinus
Keywords: Sinus Floor Augmentation; Maxillary Sinus; Bone Substitutes; Bone Regeneration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anorganic bovine bone mineral in direct sinus augmentation (Active Comparator): Anorganic bovine bone mineral
  Interventions: Procedure: Anorganic bovine bone mineral in direct sinus augmentation
- Alloplastic bone putty in direct sinus augmentation (Experimental): Alloplastic bone putty
  Interventions: Procedure: Calcium phosphosilicate alloplastic bone putty in direct sinus augmentation

INTERVENTIONS:
Procedure: Calcium phosphosilicate alloplastic bone putty in direct sinus augmentation
  Arms: Alloplastic bone putty in direct sinus augmentation
Procedure: Anorganic bovine bone mineral in direct sinus augmentation
  Arms: Anorganic bovine bone mineral in direct sinus augmentation

SUMMARY:
The purpose of this split-mouth clinical study is to evaluate the clinical, radiographic and histological outcomes of lateral window sinus augmentation with a bovine xenograft or a CPS putty bone substitute in posterior maxillary sites and the survival of implants placed in these sites following healing.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with non-contributory medical history that will present for bilateral sinus lift surgery prior to implant placement

Exclusion Criteria:

* Patients that will not agree to participate in this study or sign the consent form
* More than 8mm of residual bone height at the implant site
* Subjects smoking more than 10 cigarettes per day
* History of acute sinus infection
* History of prior maxillary sinus surgery (Caldwell-Luc, direct or indirect sinus lift, etc)
* Medications that affect bone healing (chronic steroid regimen, oral or IV bisphosphonates, etc.)
* Patients allergic to bovine derivatives
* Patients who are a carrier of transmissible disease(s) that may unnecessarily expose laboratory personnel to risks
* Females during pregnancy or lactation or females that plan to become pregnant in the following year (pregnancy test prior to enrollment)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Percentage of new bone growth in the maxillary sinus | 7 months(plus minus 1 month)
  Difference between the percentage of new bone growth between the two groups as determined by histomorphometric analysis of bone cores retrieved during implant placement surgery.

SECONDARY OUTCOMES:
Gain in vertical bone height | 6 months (plus or minus 1month)
  Patients will be seen for radiographic evaluation post-sinus surgery. A cone beam computed tomography (CBCT) will be obtained and a blinded investigator will evaluate the vertical bone height at the sites.
Radiographic bone density | 6 months (plus or minus 1 month)
  Patients will be seen for radiographic evaluation. A cone beam computed tomography(CBCT) will be obtained and a blinded investigator will evaluate the volumetric grey values at each site as an index of bone quality.
Primary implant stability | 7 months (plus or minus 1 month)
  Primary stability of implants placed in the augmented sinuses will be evaluated as a clinical index of bone density.
Marginal bone level maintenance | 12 months(plus or minus 1 month)
  Intraoral radiographs, using a paralleling technique, with customized film holders will be obtained at baseline (time of abutment connection) and at the 12-month follow-up visit and evaluated by an independent investigator to assess marginal bone levels around the implant platform. The measurements will be performed mesially and distally of each implant.

OTHER OUTCOMES:
Implant success | 2nd stage, 6&12 months post-loading
  Patients will be evaluated for clinical symptoms and implant success using predetermined criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Georgios A Kotsakis, DDS, Principal Investigator — University of Minnesota; James E Hinrichs, DDS, MS, Study Director — University of Minnesota
Locations (1):
- Advanced Education in Periodontology Clinic, Dental School, University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Hallman M, Sennerby L, Lundgren S. A clinical and histologic evaluation of implant integration in the posterior maxilla after sinus floor augmentation with autogenous bone, bovine hydroxyapatite, or a 20:80 mixture. Int J Oral Maxillofac Implants. 2002 Sep-Oct;17(5):635-43. PMID 12381063
- [Background] Del Fabbro M, Testori T, Francetti L, Weinstein R. Systematic review of survival rates for implants placed in the grafted maxillary sinus. Int J Periodontics Restorative Dent. 2004 Dec;24(6):565-77. PMID 15626319
- [Background] Mahesh L, Venkataraman N, Shukla S, Prasad H, Kotsakis GA. Alveolar ridge preservation with the socket-plug technique utilizing an alloplastic putty bone substitute or a particulate xenograft: a histological pilot study. J Oral Implantol. 2015 Apr;41(2):178-83. doi: 10.1563/AAID-JOI-D-13-00025. Epub 2013 Jun 17. PMID 23772806